CLINICAL TRIAL: NCT01424748
Title: A Single Centre, Double-blind, Three Dose Level, Parallel Group, Placebo Controlled Safety Study With Tahitian Noni Juice in Healthy Subjects
Brief Title: Clinical Trial of Tahitian Noni Juice Safety
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tahitian Noni International, Inc. (Industry)
Collaborators: TNO-BIBRA (Unknown)
Responsible Party: Brett West, Tahitian Noni Intl.
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: BIBRA5124
Record Dates: First submitted 2011-02-23; First posted 2011-08-29 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Healthy
Keywords: Noni juice; Safety

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo juice
  Interventions: Dietary Supplement: Placebo
- 30 mL Tahitian Noni Juice (Experimental): 30 mL Tahitian Noni Juice per day dose
  Interventions: Dietary Supplement: Tahitian Noni Juice
- 300 mL Tahitian Noni Juice (Experimental): 300 mL Tahitian Noni Juice per day
  Interventions: Dietary Supplement: Tahitian Noni Juice
- 750 mL Tahitian Noni Juice (Experimental): 750 mL Tahitian Noni Juice per day
  Interventions: Dietary Supplement: Tahitian Noni Juice

INTERVENTIONS:
Dietary Supplement: Tahitian Noni Juice — noni fruit juice
  Arms: 30 mL Tahitian Noni Juice; 300 mL Tahitian Noni Juice; 750 mL Tahitian Noni Juice
Dietary Supplement: Placebo — Placebo juice
  Arms: Placebo

SUMMARY:
For 28 days, healthy volunteers will consume one of four daily quantities of Tahitian Noni juice: 0 mL (placebo), 30 mL, 300 mL, or 750 mL. Hematology, biochemistry, urinalysis, vital signs, and adverse events measurements will be made at 0 (baseline), 2, and 4 weeks, as well as during a two-week follow up (week 6). Electrocardiogram (ECG) measurements will also be made for each volunteer during the pre-study screen and at week 6.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were male or female, aged between 18 and 65 years inclusive.
* Subjects had a BMI of between 19 and 30 kg/m2 inclusive.
* Prior to study commencement, subjects signed and dated a witnessed informed consent form.
* Subjects had a satisfactory documented medical history during the 21 days prior to study commencement.
* Normal blood biochemistry, haematology, urinalysis and ECG were confirmed during the 21 days prior to study commencement.
* Subjects had negative virology profile (hepatitis B surface-antigen and hepatitis C virus antibody) confirmed during the 21 days prior to study commencement.
* Females of child-bearing potential had a documented negative urine pregnancy test and were not lactating or trying to become pregnant during the course of the study. They were using an adequate method of contraception. A female of non-childbearing potential was defined as one who had been post-menopausal for at least 12 months, had been surgically sterilised, or had a hysterectomy at least 3 months prior to study start.

Exclusion Criteria:

* Subjects with any evidence or history of clinically significant hepatic or renal disorder, cardiovascular, respiratory, metabolic, immunological, neurological, psychiatric or gastrointestinal disease.
* Subjects with a history of asthma or allergic skin rash or other relevant allergic reaction.
* Subjects with known hypersensitivity or intolerance to drugs in general.
* Subjects with a history of alcohol abuse (more than 28 units per week for males and more than 21 units for females).
* Subjects who tested positive for hepatitis B surface-antigen and hepatitis C virus antibody.
* Subjects who had been on a course of prescribed drug treatment within 28 days of the study start that had not been approved by the Principal Investigator.
* Subjects who had taken any over the counter (OTC) drugs, vitamins, herbal remedies or used topically applied preparations within one week of study start unless the Principal Investigator had given approval.
* Subjects who smoked more than five cigarettes daily.
* Subjects who participated in a clinical trial or donated more than 500 ml of blood in the three months prior to study commencement.
* Female subjects who were pregnant, lactating or trying to become pregnant during the course of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2003-04; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Safety | 6 weeks
  Adverse events, electrocardiograms, vital signs, and clincial laboratory measurements recorded on day 0, 2 weeks, 4 weeks, and 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Mugglestone, MD, Principal Investigator — TNO-BIBRA